CLINICAL TRIAL: NCT04628637
Title: High GRP78 Levels in Covid-19 Infection: A Case-Control Study
Status: Completed | Type: Observational
Sponsor: Kafkas University (Other)
Collaborators: Pamukkale University Faculty of Medicine (Unknown); Acibadem Mehmet Ali Aydinlar University Faculty of Medicine (Unknown)
Responsible Party: Principal Investigator, Ramazan Sbirli, Dr., Kafkas University
Other Study IDs: Clinical-2
Record Dates: First submitted 2020-11-10; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Endoplasmic Reticulum Stress
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: Inclusion Criterias are consisted of; Not to have known acute, subacute or chronic disease history, Not to suffer from any infection in the last fortnight, Not to be on a particular medication, Presenting to the ED with reasons other than infectious complaints, and Giving their written consent to participate in the study.
  The exclusion criteria consisted of; Diagnosis of kidney and liver failure, Acute pulmonary embolism Chronic inflammatory disease history (rheumatological disease, autoimmune disease) Pregnancy Presence of any cancer diagnosis Chronic obstructive pulmonary disease Asthma disease History of cerebrovascular disease
  Interventions: Other: Serum protein level analysis
- Covid-19 (-) Pneumonia Group: Inclusion Criterias are consisted of; Presenting to the Covid-19 outpatient policlinic of the ED with pneumonia symptoms To have CT imagings were not compatible with Covid-19 pneumonia in accordance with the Radiological Society of North America Expert Consensus (RSNAEC) criteria To have nasopharyngeal swab samples taken in the ED were negative for PCR, and To give their informed consent to participate in the study. Exclusion Criteria The exclusion criteria consisted of diagnosis of kidney and liver failure, Acute pulmonary embolism Chronic inflammatory disease history (rheumatological disease, autoimmune disease) Pregnancy Presence of any cancer diagnosis Chronic obstructive pulmonary disease Asthma disease History of cerebrovascular disease To have a CT imagings that is compatible with Covid-19 pneumonia but whose PCR tests were negative
  Interventions: Other: Serum protein level analysis
- Covid-19 Infection Group: This cohort included the patients InculUsion Criteria Presenting Whose CT imagings were normal in accordance with the RSNAEC criteria and whose PCR tests were positive To have Covid-19 PCR tests were positive as a result of contact tracing, Presenting to the ED for further examination.
  The exclusion criteria consisted of; Diagnosis of kidney and liver failure, Acute pulmonary embolism Chronic inflammatory disease history (rheumatological disease, autoimmune disease) Pregnancy Presence of any cancer diagnosis Chronic obstructive pulmonary disease Asthma disease History of cerebrovascular disease To have a CT imagings that is compatible with Covid-19 pneumonia but whose PCR tests were negative.
  Interventions: Other: Serum protein level analysis

INTERVENTIONS:
Other: Serum protein level analysis — Serum GRP78 levels of the subjects were measured through a commercially available enzyme-linked immunosorbent assay (ELISA) kit (Human Glucose Regulated Protein 78 (GRP78) ELISA Kit, Sun Long, SL2048Hu, China), as per the manufacturer's protocol. The detection rate of this kit is 16 pg/mL.

SUMMARY:
Covid-19 infection was declared a global pandemic by WHO on March 11, 2020. GRP78 protein is known to be involved in the intrusion of numerous viruses. Our current study tries to provide some insight into the variation of GRP78 protein levels in patients with Covid-19(-) pneumonia, Covid-19(+) pneumonia, and CT negative Covid-19 infection in comparison to the normal population through a larger number of cases.

42 patients who have Covid-19(-) pneumonia; 72 patients who have Covid-19 infection (30 pneumonia,42 CT negative patients) and 30 patient who have no known diseases (control group) will be included in the study after the clinical and radiological evaluation. Serum GRP78 levels of the subjects will be measured through a commercially available enzyme-linked immunosorbent assay (ELISA) kit.

DETAILED DESCRIPTION:
Caused by a new type of coronavirus (SARS-CoV-2) that emerged in China in late 2019 and then were imported throughout the world, Covid-19 infection was declared a global pandemic by WHO on March 11, 2020 (1). Covid-19 infection may manifest itself in severe clinical conditions, ranging from viral upper respiratory tract infection to pneumonia, sepsis, septic shock, and even acute respiratory distress syndrome (ARDS), in symptomatic patients .

This study tries to provide some insight into the variation of GRP78 protein levels in patients with Covid-19 (-) pneumonia, Covid-19 (+) pneumonia, and CT negative Covid-19 infection in comparison to the normal population through a larger number of cases.

The present study is a prospective case-control study, and the required approval was obtained from the Ethics Committee of Pamukkale University prior to the study (60116787-020 / 26598 numbered).

The present study will be included the patients who were admitted between April 2020 and June 2020 to Covid-19 pandemic outpatient clinic of the emergency department (ED) with symptoms of upper respiratory tract infection and pneumonia, were asymptomatic, were established to be Covid-19 PCR (+) during contact tracing, and presented to the ED for further examination and treatment. After the required information concerning the study will be provided both to the patient group and to the healthy control group, the written consent forms will be obtained from all the subjects who agreed to participate in the study. The healthy volunteers with no known chronic or acute disease or drug use as well as no recent history of infection will be included study as the control group. Once these subjects will be assessed in accordance with the inclusion and exclusion criteria, they will be divided into three groups as the Covid-19(-) pneumonia group, the Covid-19 infection group, and the healthy control group.

Chest CT will performed at the time of admission of the patients to the ED was assessed under the criteria of the Radiological Society of North America Expert Consensus by an emergency physician who followed up the patient clinically. The pneumonia cases will be classified in line with these criteria and recorded in the clinical classification dataset.

Complete blood count, C-reactive protein (CRP), creatinine, urea, d-dimer, and ferritin parameters, which are routinely checked during admission to the ED, will be recorded in the dataset. For GRP78 level measurement, after 3 cc blood sample will be taken into a dry tube and centrifuged at 4000 rpm for 10 minutes, its serum section was separated, and the GRP78 level will be analyzed by the Enzyme-Linked Immunosorbent Assay (ELISA) method. In the control group, on the other hand, after 3 cc of blood was drawn into a dry tube, and another 3 cc of blood will be placed into an EDTA tube, the GRP78 level was analyzed through the same methods in the same laboratory.

Serum GRP78 levels of the subjects will be measured through a commercially available enzyme-linked immunosorbent assay (ELISA) kit (Human Glucose Regulated Protein 78 (GRP78) ELISA Kit, Sun Long, SL2048Hu, China), as per the manufacturer's protocol.

As a result of the power analysis made in line with the presumptions since a similarly-organized reference study did not exist, at least 84 people (min. 28 for each cohort) were needed to achieve 90% power at 95% confidence interval, assuming that the projected effect size would be medium-high (f = 0.4).

42 patients were eventually will be included in the Covid-19 (-) pneumonia group.

A total of 72 patients (30 Covid-19 pneumonia; 42 CT-negative Covid-19 infection) will be included in the Covid-19 infection group.

ELIGIBILITY:
Healthy group (Control group) Inclusion Criteria

* To have no known acute, subacute or chronic disease history,
* Not to not suffer from any infection in the last fortnight,
* Not to be on a particular medication
* Presenting to the ED with reasons other than infectious complaints .Giving their written consent to participate in the study.

Exclusion Criteria:

* Diagnosis of kidney and liver failure,
* Acute pulmonary embolism,
* Chronic inflammatory disease history (rheumatological disease, autoimmune disease),
* Pregnancy,
* Presence of any cancer diagnosis,
* Chronic obstructive pulmonary disease,
* Asthma disease
* History of cerebrovascular disease

Patient Groups;

Covid-19 infection Group;

Inculusion Criteria .Presenting Whose CT imagings were normal in accordance with the RSNAEC criteria.

* To have positive Covid-19 PCR test
* To have Covid-19 PCR tests were positive as a result of contact tracing,
* Presenting to the ED for further examination.

Exclusion Criteria

* Diagnosis of kidney and liver failure,
* Acute pulmonary embolism
* Chronic inflammatory disease history (rheumatological disease, autoimmune disease)
* Pregnancy
* Presence of any cancer diagnosis
* Chronic obstructive pulmonary disease
* Asthma disease
* History of cerebrovascular disease .To have a CT imagings that is compatible with Covid-19 pneumonia but whose PCR tests were negative.

Covid-19 Pneumonia Group

Inclusion Criteria

* Presenting to the Covid-19 outpatient policlinic of the ED with pneumonia symptoms
* To have CT imagings were not compatible with Covid-19 pneumonia in accordance with the .Radiological Society of North America Expert Consensus (RSNAEC) criteria
* To have nasopharyngeal swab samples taken in the ED were negative for PCR, and .To give their informed consent to participate in the study.

Exclusion Criteria

* To have diagnosis of kidney and liver failure,
* Acute pulmonary embolism
* Chronic inflammatory disease history (rheumatological disease, autoimmune disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The present study included the patients who were admitted between April 2020 and June 2020 to Covid-19 pandemic outpatient clinic of the emergency department (ED) with symptoms of upper respiratory tract infection and pneumonia, were asymptomatic, were established to be Covid-19 PCR (+) during contact tracing, and presented to the ED for further examination and treatment. After the required information concerning the study was provided both to the patient group and to the healthy control group, the written consent forms were obtained from all the subjects who agreed to participate in the study. The healthy volunteers with no known chronic or acute disease or drug use as well as no recent history of infection were included study as the control group. Once these subjects were assessed in accordance with the inclusion and exclusion criteria, they were divided into three groups as the Covid-19(-) pneumonia group, the Covid-19 infection group, and the healthy control group.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Determination of the change of the serum GRP-78 protein levels in patients who have Covid-19 infection compared to control group | 2 months
  The change of the serum levels of the GRP-78 protein levels in patient who have Covid 19 infection compared to control group. It will be determined whether GRP-78 protein level change in Covid-19 infection.
Determination of the change of the serum GRP-78 protein levels in patients who have Covid-19 infection compared to Covid-19 negative pneumonia group. | 2 months
  The change of the serum levels of the GRP-78 protein levels in patient who have Covid 19 infection compared to Covid-19 negative pneumonia group.. It will be determined whether GRP-78 protein level change in Covid-19 (-) pneumonia.

SECONDARY OUTCOMES:
Determination of the correlations between laboratory parameters, clinical parameters and radiological parameters | 2 months
  Correlationships will be analysed between Complete blood count, C-reactive protein (CRP), creatinine, urea, d-dimer, and ferritin parameters, CURB-65 score, PORT score, symptom duration, CT severity score.

CONTACTS AND LOCATIONS:
Locations (1):
- Aylin Koseler, Denizli, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to share IPD.